CLINICAL TRIAL: NCT03213327
Title: StayOK - an Innovative Measuring Instrument for the Early Identification and Treatment of Psychosocial Risks
Acronym: StayOK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Collaborators: Health and Medical Services (Unknown); Helsana (Unknown); Neomentum (Unknown); Sanatorium Kilchberg AG (Other); Design your life (Unknown)
Responsible Party: Principal Investigator, Aureliano Crameri, Dr. phil., Zurich University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BASEC-Nr. 2016-00879
Record Dates: First submitted 2017-06-15; First posted 2017-07-11 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Mental Health Disorder
Keywords: mental health; assessment; health promotion; case management; health insurance
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Patients are examined at two time points: baseline and 12 weeks after the Intervention.
  The Intervention consists of health-promoting advices provided by the software algorithm. The effect of this intervention is evaluated 12 weeks after.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case management (Other): Case management program Utilization of the StayOk web application
  Interventions: Device: StayOk web application

INTERVENTIONS:
Device: StayOk web application — Patients fill in the questionnaires of the web application and receive an analyzed profile of their psychosocial condition and health-promoting advices

SUMMARY:
The validity and the sensitivity of different measures implemented in the web application StayOk are investigated. The measures are used primarily for the assessment and the early identification of psychosocial risks. Secondarily, the results of the assessment are applied to generate health-promoting advices for the user of the web application.

ELIGIBILITY:
Inclusion Criteria:

* at 16 years of age
* mild to moderate psychological distress

Exclusion Criteria:

* serious cognitive impairment due to dementia or cerebrovascular insult
* Insufficient knowledge of one of the following languages: German, French, Italian or English

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Psychological distress | 0 week (first assessment)
  The psychological distress is assessed by the Brief Symptom Inventory (BSI; Derogatis & Melisaratos, 1983)
Work-related sense of coherence | 0 weeks
  The work-related sense of coherence is assessed by the Work Sense of Coherence (W-SoC 9; Jenny et al., 2016)
Perceived self-efficacy | 0 weeks
  This aspect is measure by the General Self-Efficacy Scale (GSE; Damásio et al., 2016)

SECONDARY OUTCOMES:
Effectiveness of health-promoting advices | 12 weeks after the first assessment
  The effectiveness of the advices generated by the software is assessed by means of a self-developed questionnaire: Participants are inquired as to (1) whether they put in practice the advices and (2) how they evaluate the benefit of the applied advices and the consequent satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes von Wyl, Prof, Principal Investigator — Zurich University of Applied Sciences
Locations (1):
- Helsana, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Jenny GJ, Bauer GF, Vinje HF, Vogt K, Torp S. The Application of Salutogenesis to Work. 2016 Sep 3. In: Mittelmark MB, Sagy S, Eriksson M, Bauer GF, Pelikan JM, Lindstrom B, Espnes GA, editors. The Handbook of Salutogenesis [Internet]. Cham (CH): Springer; 2017. Chapter 20. Available from http://www.ncbi.nlm.nih.gov/books/NBK435821/ PMID 28590629
- [Background] Damasio BF, Valentini F, Nunes-Rodriguez SI, Kliem S, Koller SH, Hinz A, Brahler E, Finck C, Zenger M. Is the General Self-Efficacy Scale a Reliable Measure to be used in Cross-Cultural Studies? Results from Brazil, Germany and Colombia. Span J Psychol. 2016 May 26;19:E29. doi: 10.1017/sjp.2016.30. PMID 27225231
- See also: Stay OK — https://www.zhaw.ch/en/psychology/research/clinical-psychology-and-health-psychology/prevention-and-health-promotion/stay-ok/